CLINICAL TRIAL: NCT01352806
Title: Identification of the Lumbar Interspinous Spaces; Palpation Versus Ultrasound Versus Fluoroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Saifi fayez, Hadassah Medical Orginization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 039910-HMO-CTIL
Record Dates: First submitted 2011-04-27; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-04

CONDITIONS: Accuracy of Identifying the Intralaminar Space
Keywords: accuracy of identifying intralaminar space

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fluoroscopy, palpation, ultrasound (Experimental): in the same subject we will compare the accuracy of identifying the intralaminar space by three technique, fluoroscopy, ultrasound, palpation.
  Interventions: Procedure: identification of the lumbar interspinous space using fluoroscopy versus ultrasound versuspalpation

INTERVENTIONS:
Procedure: identification of the lumbar interspinous space using fluoroscopy versus ultrasound versuspalpation — Copmarison of multiple technique for identification of the lumbar interspinous space,which is fluoroscopy,ultrasound and palpation

SUMMARY:
The of epidurals and spinals, relies primarily on palpation of anatomic landmarks that are not always easy to find, More so, even after correct identification of palpable landmarks, Variability exists leading to performing neuraxial injection in undetermined intralaminar level. The most accurate method for identifying the interspace is the using of the fluoroscopy or CT technique, but exposure to radiation and availability make it unpractical in majority of cases. As ultrasound technology becomes more accessible to the clinician, it holds great potential to facilitate performing neuraxial anesthesia by the anesthesiologist in routine cases.

The aim of this study to compare the accuracy of identifying the intervertebral space, between manual palpation, versus ultrasound versus fluoroscopy.

DETAILED DESCRIPTION:
Neuraxial anesthesia relies upon a sound knowledge of anatomy to accurately direct needle placement both to achieve consistent success, and to avoid damage to other nearby structures. This prospective randomized study, will be performed in the pain management unit. We will assess patients who are scheduled to receive an epidural steroid injection. The investigator will request permission fro the ethics committee of Hadassah Medical Hospital.

Three anesthesiologist will perform this study, every one of the anesthesiologist will be asked to identify intralaminar space by one technique and we will compare the accuracy of the identifying of the intralaminar space.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for epidural steroid injection under fluoroscopy technique.
* Age above 18 years

Exclusion Criteria:

* Inability to understand consent form.
* refusing to sign the consent form.
* contraindication for neuraxial injection.
* local or systemic infection.
* pregnant women.
* previous spine surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of identifying the intralaminar space | one year

SECONDARY OUTCOMES:
Patient satisfaction | one year

CONTACTS AND LOCATIONS:
Overall Officials: Fayez Saifi, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel